CLINICAL TRIAL: NCT03660150
Title: Evaluation of Long-term Health-related Quality of Life After Massive Burn Injury : A Twenty Years' Experience in a Burn Center
Brief Title: Health-related Quality of Life After Massive Burn Injury
Acronym: HR - QOL MR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2018_003
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Patients With Massive Burn Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of health-related quality of life — Short Form-36 Medical Outcomes Survey (SF-36), and Brief Version of Burn Speciﬁc Health Scale (BSHS-B) are used for the present evaluation.

SUMMARY:
Massive burns are serious life-threatening conditions. Recent advances in their management now allow the survival of a growing number of patients. The burn care paradigm is transformed: the evaluation of survival at the end of acute care is no longer sufficient for a good evaluation of practices; the attention now focuses on long-term health-related quality of life (HR-QOL).The recently validated French translation of the burn specific health scale brief version makes this evaluation now feasible in French burn centers. The objectives of this study are to evaluate the HR-QOL of massive burn survivors, to compare it to another chronic condition (necrotizing fasciitis) and to determine the main predictive factor of health-related quality of life. This study is retrospectively conducted in 18 patients who survived a massive burn injury involving more than 80% of the total body surface area, or more than 70% of the total body surface area if the injury occured during childhood and who were treated between 1997 and 2017 in our Lyon burn center. Short Form-36 Medical Outcomes Survey (SF-36), and Brief Version of Burn Speciﬁc Health Scale (BSHS-B) are used for the present evaluation.

DETAILED DESCRIPTION:
The hypotheses are as follows:

* the HR-QOL of massive burns shows a significative alteration compared to general population
* this alteration is comparable with another chronic disease
* the main predictors of impaired quality of life related to physical health status are hand injury, age at time of burn and time since burn
* the main predictive factors of change in quality of life related to mental health status are age of onset and facial involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 14 years of age
2. Patients with a childhood burn reaching more than 70% of the total body surface OR Adult patients with burns of more than 80% of total body surface area
3. Patients who were treated at the burn center between January 1997 and January 2017
4. Patients who survived after initial hospitalization for burn management

Exclusion Criteria:

1. Patients with superficial burning, without sequelae or with extensive sequelae at less than 70% of total body surface area in children and less than 80% of total body surface area in adults
2. Patients who expressed opposition to their participation in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Survivors of a massive burn injury involving more than 80% total body surface area, or more than 70% of the total body surface area if the injury occured during childhood and who were treated between 1997 and 2017 in a Lyon burn center
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Short Form-36 Medical Outcomes Survey (SF-36) sub domain score | Data concerning HR-QOL was retrospectively collected in July 2018 for all patients with a massive burn injury occuring during 1997 and 2017
  The impact of massive burn injury is measured for each SF 36 sub domain and compared to general population score.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Braye, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Croix-Rousse Hospital, Lyon, France

IPD SHARING:
Plan to Share IPD: No